CLINICAL TRIAL: NCT01513447
Title: Intracutaneous Sterile Water Injection as an Adjunct to Neuraxial Labor Analgesia: A Randomized Controlled Trial
Brief Title: Intracutaneous Sterile Water Injections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low qualified candidate enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00057039
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Labor Pain
Keywords: sterile water injections; back labor
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sterile Water Injection (Active Comparator): In the sitting position, study subjects will receive a total of 0.4 mL of "study drug" via four intracutaneous injections: bilateral injections at the posterior superior iliac spine and bilateral injections at 1 cm medial and 1-2 cm inferior to the first point.
  Interventions: Drug: Intracutaneous injections
- Normal Saline Injection (Placebo Comparator): In the sitting position, study subjects will receive a total of 0.4 mL of "study drug" via four intracutaneous injections: bilateral injections at the posterior superior iliac spine and bilateral injections at 1 cm medial and 1-2 cm inferior to the first point.
  Interventions: Drug: Intracutaneous injections

INTERVENTIONS:
Drug: Intracutaneous injections — Four intracutaneous injections: two sites lateral to the lumbosacral spine and two sites 2-3 centimeters below and 1- 2 centimeters medial to the original two injections sites. 0.1 millimeters of the study drug is injected between the dermal layers at each of the four sites. The injections are administered sequentially, with the series of four injections, performed two at a time, completed in 20-30 seconds.

SUMMARY:
For most women, the most significant pain they will experience is the pain associated with childbirth. Up to one-third of women experience "back labor", this typically occurs when the fetus assumes varying degrees of malposition, especially the occiput posterior position, and causes additional constant pressure against the maternal spine and pelvis. "Back labor" presents as constant pain, that occurs even between contractions. It is often difficult to manage, by the patient, the obstetrician, and the anesthesiologist, and may increase the rate of instrumental and caesarian delivery.

Epidural anesthesia/analgesia is the most common and effective intervention used to help women cope with labor pain. Dilute concentrations of local anesthetic and opioid provide complete analgesia for most women. Some women, however, have breakthrough pain, often due to "back labor," and require more concentrated drug solutions. This increases the side effects associated with these drugs (e.g., hypotension, pruritus, motor block), thus treatment of this pain poses a challenge for the anesthesiologist and the obstetrician.

Sterile water injections (SWI) are a simple and well-established method of managing labor pain among midwives. This intervention was first used to alleviate pain associated with kidney stones, and was introduced to obstetrics in the 1970s. Using a syringe, small amounts of sterile water is deposited subcutaneously near the sacral area. The sterile water causes osmotic and mechanical irritation resulting in a brief (15-30 second) and significant stinging sensation. The onset of pain relief follows almost immediately and may last for up to two hours. The procedure can be repeated a number of times.

Sterile water for pain management is most often administered using four intracutaneous injections: two sites lateral to the lumbosacral spine and two sites 2-3 cm below and 1-2 cm medial to the original two injection sites. 0.1 mL of sterile water is injected between the dermal layers to raise a small bleb on the skin surface at each of the four sites. In labor, the injections are administered sequentially during a uterine contraction, with the series of four injections, performed two at a time, completed within 20-30 seconds.

The investigators hypothesize that the use of sterile water injections in women with neuraxial analgesia with breakthrough pain will result in decreased local anesthetic requirements and increase patient satisfaction.

DETAILED DESCRIPTION:
Since it is assumed that the neuraxial anesthetic is placed prior to transition to active phase of labor, the patient will receive the intervention when they report breakthrough pain. Prior to administration of the intervention, the adequacy of the existing neuraxial anesthetic will be verified as bilateral decreased discrimination to cold from T8 to the sacrum. Four tuberculin syringes, each containing 0.1 mL of the assigned solution labeled "study drug" will be prepared. Patients allocated to the study group will receive sterile water, and those allocated to the control group will receive sterile normal saline solution.

The area to be injected will be prepared with chlorhexidine wipes to ensure sterility. In the sitting position, study subjects will receive a total of 0.4 mL of "study drug" via four injections: bilateral injections at the posterior superior iliac spine on and bilateral injections at 1 cm medial and 1-2 cm inferior to the first point.

Patients will be asked to rate their overall labor pain using a 0-100 mm visual analog scale (VAS) for pain prior to study drug administration and every 30 minutes until commencement of pushing. They will also be asked to specifically rate low back pain with the VAS. Analgesia administration data from the time of study drug injection, including maintenance epidural solution volume, time of first patient controlled epidural analgesia (PCEA) bolus request, number of PCEA bolus requests and delivered doses, total PCEA bupivacaine dose, time to first request for manual rebolus, number of manual bolus doses, manual bolus bupivacaine dose, total bupivacaine dose and total fentanyl dose.

Additional recorded data will include maternal age, height, weight, cervical dilation at initiation of neuraxial analgesia and at study drug administration, duration of labor (initiation of analgesia to delivery), maximum oxytocin infusion rate during labor, and mode of delivery. A "total labor pain score" will be assessed approximately 60 minute after delivery, as well as satisfaction with labor analgesia using a 100-mm VAS.

ELIGIBILITY:
Inclusion Criteria:

* multiparous women
* spontaneous labor
* at least 18 years of age
* presenting for vaginal delivery with cervical dilation of 4 centimeters or less

Exclusion Criteria:

* nulliparous
* less than 18 years old
* contraindication to placement of neuraxial anesthetic
* skin infection in area to be injected
* medical therapies considered to result in tolerance to opioids
* history of chronic pain (requiring regular medical follow-up with pain specialists)
* recent use of opioid analgesics (within the year preceding pregnancy)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Wong, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Creehan PA. Pain relief and comfort measures in labor. In: Simpson KR, Creehan PA, editors. AWHONN's Perinatal Nursing, 3rd edn. Philadelphia, PA: Lippincott Williams & Wilkins; 2008. pp. 444-72.
- [Background] Cervero F, Tattersall JE. Somatic and visceral sensory integration in the thoracic spinal cord. Prog Brain Res. 1986;67:189-205. doi: 10.1016/s0079-6123(08)62763-6. No abstract available. PMID 3823471
- [Background] Bengtsson J, Worning AM, Gertz J, Struckmann J, Bonnesen T, Palludan H, Olsen PR, Frimodt-Moller C. [Pain due to urolithiasis treated by intracutaneous injection of sterile water. A clinically controlled double-blind study]. Ugeskr Laeger. 1981 Dec 14;143(51):3463-5. No abstract available. Danish. PMID 7039061
- [Background] Odent M. [Letter: Lumbar reflexotherapy. Efficacy in the treatment of nephrotic colic and in obstretrical analgesia]. Nouv Presse Med. 1975 Jan 18;4(3):188. No abstract available. French. PMID 1129076
- [Background] Huntley AL, Coon JT, Ernst E. Complementary and alternative medicine for labor pain: a systematic review. Am J Obstet Gynecol. 2004 Jul;191(1):36-44. doi: 10.1016/j.ajog.2003.12.008. PMID 15295342
- [Background] Reynolds JL. Intracutaneous sterile water for back pain in labour. Can Fam Physician. 1994 Oct;40:1785-8, 1791-2. PMID 7950471
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Martensson L, McSwiggin M, Mercer JS. US midwives' knowledge and use of sterile water injections for labor pain. J Midwifery Womens Health. 2008 Mar-Apr;53(2):115-22. doi: 10.1016/j.jmwh.2007.09.008. PMID 18308260
- [Background] Hutton EK, Kasperink M, Rutten M, Reitsma A, Wainman B. Sterile water injection for labour pain: a systematic review and meta-analysis of randomised controlled trials. BJOG. 2009 Aug;116(9):1158-66. doi: 10.1111/j.1471-0528.2009.02221.x. Epub 2009 May 14. PMID 19459860
- [Background] Wong CA, McCarthy RJ, Hewlett B. The effect of manipulation of the programmed intermittent bolus time interval and injection volume on total drug use for labor epidural analgesia: a randomized controlled trial. Anesth Analg. 2011 Apr;112(4):904-11. doi: 10.1213/ANE.0b013e31820e7c2f. PMID 21430035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 4/17/2012, ended 10/26/2012. Recruitment stopped due to low number of subjects meeting study criteria for entry.
Pre-assignment Details: Delivery of infant in less than 90 minutes from recruitment.
Period: Overall Study
Arm/Group | Sterile Water Injection | Normal Saline Injection
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Laboring women requesting labor analgesia
Groups:
- Total: Total of all reporting groups
Arm/Group | Sterile Water Injection | Normal Saline Injection | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (10) | 31 (4) | 31 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Breakthrough Back Labor Pain
Description: It is anticipated that intracutaneous sterile water injections will provide additional pain relief as part of a multimodal analgesic regimen in women, especially in women with back labor.
Time Frame: within 24 hours
Measure: Number; unit: participants
Arm/Group | Sterile Water Injection | Normal Saline Injection
Number analyzed (Participants) | 3 | 5
participants | 0 | 2
Statistical Analysis 1: Comparison: Sterile Water Injection vs Normal Saline Injection; Test type: Superiority or Other; p = 0.67, Fisher Exact

2. Secondary Outcome: Total Local Anesthetic Consumption
Description: It is anticipated that intracutaneous sterile water injections will decrease the amount of local anesthetic consumption.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Sterile Water Injection | Normal Saline Injection
Number analyzed (Participants) | 3 | 5
milliliters | 190 (104) | 234 (60)
Statistical Analysis 1: Comparison: Sterile Water Injection vs Normal Saline Injection; Test type: Superiority or Other; p = 0.29, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 102, 95% CI 2-sided [-230 to 171]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from intervention until delivery of infant, for up to 24 hours
Arm/Group | Sterile Water Injection | Normal Saline Injection
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Subjects recruitment unsuccessful because of low number of subjects that were eligible for study inclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No